CLINICAL TRIAL: NCT01144182
Title: VALOR (Veterans Affairs Lowering Readmissions) in Heart Failure Study
Brief Title: Veterans Affairs Lowering Readmission in Heart Failure
Acronym: VALOR in HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRP 09-412
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
Keywords: heart failure; quality of life; readmissions
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current Best Practice (CBP) (No Intervention): CBP received no intervention and only current best practices for inpatient HF care.
- Quality improvement program (QIP) (Active Comparator): Comprehensive quality improvement program (QIP) intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients.
  Interventions: Behavioral: Comprehensive quality improvement program (QIP)

INTERVENTIONS:
Behavioral: Comprehensive quality improvement program (QIP) — Comprehensive quality improvement program (QIP) that intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients.
  Arms: Quality improvement program (QIP)

SUMMARY:
Heart failure (HF) greatly increases mortality and lowers quality of life (QOL). HF is the most common indication for readmission in older adults and the most frequent reason for 30-day readmission. Medications and restriction of dietary sodium constitute crucial therapy to lower HF recurrence. However, adherence to medications and dietary recommendations is low in HF patients. Nonadherence is often due to an interaction among the environment, the patient and providers. In the VALOR in Heart Failure Study, we will assess a novel quality improvement program (QIP) to improve HF care using a pretest-posttest design. This interdisciplinary theory-based prospective experimental study will target improving HF treatment using patient-based behavioral and checklist intervention, as well as provider and system-targeted checklists and treatment defaults (posttest or intervention phase); this will be compared to current best practice (CBP) evaluated in the pretest (pretest or pre-intervention) phase. It is hypothesized that the QIP, which intervenes on patient, provider and system levels, will improve QOL and lower HF recurrence compared to CBP.

DETAILED DESCRIPTION:
Heart failure (HF) greatly increases mortality and lowers quality of life (QOL). HF is the most common indication for readmission in older adults and the most frequent reason for 30-day readmission. Medications and restriction of dietary sodium constitute crucial therapy to lower HF recurrence. However, adherence to medications and dietary recommendations is low in HF patients. Nonadherence is often due to an interaction among the environment, the patient and providers. In the VALOR in Heart Failure Study, we will assess a novel quality improvement program (QIP) to improve HF care using a pretest-posttest design. This interdisciplinary theory-based prospective experimental study will target improving HF treatment using patient-based behavioral and checklist intervention, as well as provider and system-targeted checklists and treatment defaults (posttest or intervention phase); this will be compared to current best practice (CBP) evaluated in the pretest (pretest or pre-intervention) phase. It is hypothesized that the QIP, which intervenes on patient, provider and system levels, will improve QOL and lower HF recurrence compared to CBP.

The primary specific aims are 1) To test the effect of QIP on HF-specific quality of life compared to the CBP group, and 2) To evaluate the impact of QIP group on general quality of life compared to the CBP group.

Secondary specific aims are to:

1) assess the effect of QIP on medication adherence at 3 months, 2) examine the effect of QIP on diet adherence at 3 months, and 3) evaluate the effect of QIP on satisfaction, and 4) assess the effect of QIP on intervention acceptability. We will also examine the impact of QIP at 3 months on keeping routine outpatient visits, health-care utilization, exercise capacity, weight, perceived stress, depression, cardiovascular events and deaths.

Exploratory aim is to examine the effect of the QIP on 30 day post-discharge HF readmission rates compared to CBP.

We have enrolled 136 veterans being discharged from the hospital with a diagnosis of HF. Patients enrolled in the pretest phase will receive the HF management based on current best practice (CBP). Patients enrolled in the posttest phase receive the comprehensive quality improvement program (QIP) that intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients. Data, including quality of life (QOL), medication adherence, and dietary adherence, will be collected from patients at baseline (prior to hospital discharge) and 3 months. Hospital readmissions, emergency room visits, and healthcare utilization will be tracked for 6 months. If, as expected, there are no differences in demographic or other confounders (EF, comorbidities, etc), the pretest and posttest groups will be compared by the Fisher's Exact test for discrete outcomes (30-day readmissions or ER visits). We will use the Student's ttest (two-tailed) for normally distributed outcomes and the Wilcoxon rank-sum test for categorical variables and continuous variables not normally distributed.

This study will inform and enhance quality improvement efforts in heart failure care in VA New York Harbor and elsewhere. It will also provide data for a rigorous effectiveness trial to test this promising intervention that could reduce HF recurrence and improve QOL in HF. If this promising theory-driven approach can work in a clinical setting where improvements in HF care are so urgent, it will be an important scientific contribution.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with either systolic or diastolic HF will be identified through ongoing daily prospective manual search of admission records in VA NYHHS
* Men and women ( 21 years) being discharged after a HF admission will be eligible
* They must have an available phone

Exclusion Criteria:

* Patients with poor short-term survival (< 3 months)
* recent major surgery (< 1 month)
* planned discharge to a long-term-care facility
* severe dementia or other serious psychiatric illness
* temporarily in the area
* those unable to provide consent, refusal to participate
* logistic or discretionary reasons (including participation in another study) will be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD MSc, Principal Investigator — VA New York Harbor Health Care System
Locations (1):
- VA New York Harbor Health Care System, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Quality Improvement Program (QIP): Comprehensive quality improvement program (QIP)
  Comprehensive quality improvement program (QIP): Comprehensive quality improvement program (QIP) that intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients.
Period: Overall Study
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Started | 68 | 68
Completed | 51 | 47
Not Completed | 17 | 21
Not completed — Death | 5 | 6
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Current Best Practice (CBP): Current best practice (CBP) receives the current treatment for patients discharged with heart failure
- Total: Total of all reporting groups
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP) | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75.3 [61.4 to 83.5] | 74.8 [64.7 to 84.6] | 74.8 [63.8 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 66 | 68 | 134
Race/Ethnicity, Customized [Number; unit: participants]
  White (non-Hispanic) | 37 | 30 | 67
  Black (non-Hispanic) | 14 | 16 | 30
  Hispanic | 13 | 19 | 32
  Other | 4 | 3 | 7
Marital Status [Number; unit: participants]
  Married | 15 | 18 | 33
  Not Married | 53 | 50 | 103
Education [Number; unit: participants]
  High school graduate or below | 34 | 32 | 66
  Some college or higher | 34 | 36 | 70
Employment status [Number; unit: participants]
  Employed | 6 | 4 | 10
  Not employed | 62 | 64 | 126
Campus [Number; unit: participants]
  Manhattan | 50 | 45 | 95
  Brooklyn | 18 | 23 | 41
BNP [Median (Inter-Quartile Range); unit: pg/mL] — B-type natriuretic peptide
  pg/mL | 645.0 [433.0 to 1512.5] | 739.0 [383.0 to 1702.0] | 696.0 [413.0 to 1580.0]
Number of heart failure medications [Median (Inter-Quartile Range); unit: number of heart failure medications] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
Length of hospital stay [Median (Inter-Quartile Range); unit: days] | 6 [3 to 9] | 6 [4 to 9] | 6 [3 to 9]

OUTCOME MEASURES:

1. Secondary Outcome: Standardized Mental Component Score
Description: Assesses General Quality of Life from VR-36, with scores ranging from 0 to 100 and higher score indicating better quality of life
Time Frame: 3 months after discharge
Population: 51 patients in CBP and 47 patients in QIP had a follow-up visit. However, 1 participant in each arm did not complete the VR-36, such that there are only 50 participants analyzed in CBP and 46 in QIP for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 48.8 [35.6 to 58.9] | 53.2 [39.6 to 58.5]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = .56, Wilcoxon (Mann-Whitney) — For this pilot study, significance level was set at p<0.05

2. Secondary Outcome: Physical Functioning
Description: Subscale of General Quality of Life from VR-36, with scores ranging from 0 to 100 and higher score indicating better quality of life
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 37.5 [15.0 to 60.0] | 41.4 [25.0 to 65.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Role Physical
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: 51 patients in CBP and 47 patients in QIP had a follow-up visit. However, 1 participant in each arm did not complete the VR-36. Additionally, a second participant in CBP did not complete the role physical subscale items, leaving a total of 49 in CBP and 46 in QIP for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 49 | 46
units on a scale | 50.0 [18.8 to 68.8] | 53.1 [31.3 to 87.5]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain Index
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 51.0 [31.0 to 84.0] | 61.5 [41.0 to 100.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: General Health
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 41.0 [20.0 to 57.0] | 57.0 [35.0 to 77.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Vitality
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 45.0 [30.0 to 65.0] | 50.0 [35.0 to 70.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Social Functioning
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 62.0 [37.5 to 75.0] | 75.0 [50.0 to 100.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Role Emotional
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 66.7 [33.3 to 100.0] | 75.0 [50.0 to 100.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Mental Health
Description: as for outcome 2
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 74.0 [56.0 to 88.0] | 80.0 [48.0 to 88.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney)

10. Primary Outcome: General Quality of Life From the Standardized Physical Component Score
Description: as for outcome 1
Time Frame: 3 months after discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Quality Improvement Program (QIP): Comprehensive quality improvement program (QIP)
  Comprehensive quality improvement program (QIP): Comprehensive quality improvement program (QIP) that intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients.
Arm/Group | Current Best Practice (CBP) | Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 31.6 [25.4 to 38.5] | 35.5 [28.0 to 44.3]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Physical Subscale of Heart Failure Specific Quality of Life
Description: Subscale of the Minnesota Living with Heart Failure Questionnaire (HF-specific quality of life measure). Scores range from 0-40, with higher scores indicating poorer QOL.
Time Frame: 3 months after discharge
Population: 51 patients in CBP and 47 patients in QIP had a follow-up visit. However, 1 participant in each arm did not complete the Minnesota Living with Heart Failure Questionnaire, such that there are only 50 participants analyzed in CBP and 46 in QIP for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 21.5 [8.0 to 32.0] | 19.0 [9.0 to 24.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Heart Failure Specific Quality of Life
Description: Measured by Minnesota Living with Heart Failure Questionnaire. Scores range from 0-105, with higher scores indicating poorer QOL.
Time Frame: 3 months after discharge
Population: 51 patients in CBP and 47 patients in QIP had a follow-up visit. However, 1 participant in each arm did not complete the MLHFQ, such that there are only 50 participants analyzed in CBP and 46 in QIP for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 42.5 [20.0 to 67.0] | 38.0 [21.0 to 55.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Emotional Subscale of Heart Failure Specific Quality of Life
Description: Subscale of the Minnesota Living with Heart Failure Questionnaire (HF-specific quality of life measure). Scores range from 0-25, with higher scores indicating poorer QOL.
Time Frame: 3 months after discharge
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Current Best Practice (CBP) | Comprehensive Quality Improvement Program (QIP)
Number analyzed (Participants) | 50 | 46
units on a scale | 7.0 [3.0 to 18.0] | 6.0 [3.0 to 13.0]
Statistical Analysis 1: Comparison: Current Best Practice (CBP) vs Comprehensive Quality Improvement Program (QIP); Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Quality Improvement Program (QIP): Quality improvement program (QIP)
  The comprehensive quality improvement program (QIP): Comprehensive quality improvement program (QIP) that intervenes on patient, provider and system levels. The QIP will consist of 3 monthly phone calls to promote diet and medication adherence using the transtheoretical model as a behavioral framework and checklists to facilitate patients' self-monitoring of their diet, physical activity, weight and medication taking. Further, providers during the posttest phase will use checklists for inpatient and outpatient care of HF patients.
Arm/Group | Current Best Practice (CBP) | Quality Improvement Program (QIP)
Serious Adverse Events (participants affected / at risk) | 7/68 | 8/68
Other Adverse Events (participants affected / at risk) | 6/68 | 5/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Current Best Practice (CBP) (N=68) | Quality Improvement Program (QIP) (N=68)
Death (General disorders) | 5 (5) | 6 (6)
myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Current Best Practice (CBP) (N=68) | Quality Improvement Program (QIP) (N=68)
Coronary artery bypass graft (Surgical and medical procedures) | 1 (1) | 0 (0)
angina (Cardiac disorders) | 2 (2) | 1 (1)
broken bone (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hypertensive emergency (Cardiac disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes